CLINICAL TRIAL: NCT04776967
Title: The Effect of Total Compression Time and Rate (Slope) of Compression on Incidence of Symptomatic Eustachian Tube Dysfunction and Middle Ear Barotrauma: A Phase II Prospective Study.
Brief Title: Effect of Total Compression Time and Rate (Slope) on Incidence of Symptomatic ETD and MEB: A Phase II Prospective Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Owen J O'Neill, MD, MPH, Medical Director Division of Undersea & Hyperbaric Medicine, Northwell Health
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Compression Hyperbaric II
Record Dates: First submitted 2021-02-10; First posted 2021-03-02 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Eustachian Tube Dysfunction; Middle Ear Barotrauma; Middle Ear Disease; Middle Ear; Injury; Pressure Injury; Ear Barotrauma
Keywords: Ear Pressure; Otic Barotrauma; Hyperbaric; Pressure Equalization; O'Neill Grading System; Compression Rate
MeSH Terms: conditions — Wounds and Injuries; Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Compression Profile 4 (Active Comparator): Compression Profile/Schedule 4 = 10 minute linear, Total Time Interval of Compression to treatment depth = 10 minutes, Rate (slope) of compression = Linear rate of compression = 4.5 fsw/min to arrival at treatment depth 45 fsw
  Interventions: Procedure: Hyperbaric Compression Profile
- Compression Profile 3 (Active Comparator): Compression Profile/Schedule 3 = 10 minute non-linear, Total Time Interval of Compression to treatment depth = 10 minutes Rate (slope) of compression = Non-Linear rate of compression = 3 fsw/min to a depth of 17 fsw, then 5 fsw/min up to a depth of 38.5 fsw, then 6.5 fsw/min to arrival at the treatment depth of 45 fsw
  Interventions: Procedure: Hyperbaric Compression Profile
- Compression Profile 2 (Active Comparator): Compression Profile/Schedule 2 = 15 minute linear, Total Time Interval of Compression to treatment depth = 15 minutes Rate (slope) of compression = Linear rate of compression = 4.5 fsw/min to arrival at the treatment depth 45 fsw
  Interventions: Procedure: Hyperbaric Compression Profile
- Compression Profile 1 (Active Comparator): Compression Profile/Schedule 1 = 15 minute non-linear, Total Time Interval of Compression to treatment depth = 15 minutes Rate (slope) of compression = Non-Linear rate of compression = 2 fsw/min to a depth of 13 fsw, then 3 fsw/min up to a depth of 35 fsw, then 5 fsw/min to arrival at the treatment depth of 45 fsw
  Interventions: Procedure: Hyperbaric Compression Profile

INTERVENTIONS:
Procedure: Hyperbaric Compression Profile — A total of 4 randomized hyperbaric treatment compression profiles (accepted standards of care) will be alternated over the patients course of treatment on a daily basis daily to the prescribed treatment depth.
  Other Names: Hyperbaric Compression Schedule

SUMMARY:
Eustachian tube dysfunction (ETD) and middle ear barotrauma (MEB) are common reported complications during hyperbaric oxygen treatment. The Phase I study data was the first to demonstrate a statistically significant decrease in the occurrence of symptomatic ETD and middle ear barotrauma (MEB). The Phase I Trial suggested the total time interval and rate (slope) of compression (ROC) may be a determining factor in ETD and MEB. This Phase II study investigates an optimal total time interval and rate of compression to reduce ETD and MEB when considering each multiplace treatment (with multiple patients) as the unit of observation collectively as a group, rather than for each individual patient.

Data will be collected prospectively on group patient-treatment exposures. The investigators randomly assigned patient-treatment group exposures to four different time interval and rate (slope) of compression. These total time intervals of compression and rates (slopes) of compression are identical to those used in the Phase I trial. All patients experiencing symptoms of ETD and MEB requiring compression stops will be evaluated post treatment to confirm the presence of ETD and MEB using the O'Neill Grading System (OGS). Data will be analyzed using the IBM-SPSS statistical software program.

The number of compression holds observed in each of the 4 compression schedules, similar to ther Phase I trial will be recorded. Patients who are symptomatic and require compression stops (as in the Phase I trial) using a United States Navy Treatment Table 9 (USN-TTN9) during elective hyperbaric oxygen treatments in a Class A multiplace hyperbaric chamber will be analyzed. Analysis using descriptive and inferential statistics will be applied to the patients requiring first stops in the 4 compression profiles. This Phase II study increases the sample size of treatments and they will be combined with the total number of treatments used in the original phase I study. This will increase power to facilitate detailed descriptive analysis and to determine if the findings are robust in the phase I study.

DETAILED DESCRIPTION:
Eustachian tube dysfunction (ETD) and middle ear barotrauma (MEB) are common reported complications during hyperbaric oxygen treatment. The investigators Phase I study data was the first to demonstrate a statistically significant decrease in the occurrence of symptomatic ETD and middle ear barotrauma (MEB). The Phase I Trial suggested the total time interval and rate (slope) of compression (ROC) may be a determining factor in ETD and MEB. This Phase II study investigates an optimal rate of compression to reduce ETD and MEB when considering each multiplace treatment (with multiple patients) as the unit of observation as a group, rather than for each individual patient.

Data will be collected prospectively on group patient-treatment exposures. The investigators will randomly assign patient-treatment group exposures to four different time interval and rate (slope) of compression. All patients, within every patient-treatment group exposure, received all 4 compression profiles (CP) on a rotating basis, in effect having patients serve as their own controls in a crossover design and to reduce the risk of treatment order on the effects observed. These compression rates and slopes were identical to those used in the Phase I trial. All patients experiencing symptoms of MEB requiring compression stops will be evaluated post-treatment for the presence of ETD and MEB using the O'Neill Grading System (OGS) for ETD/MEB.

For approximately 10 years, the investigators hyperbaric center used a routine daily multiplace chamber treatment protocol to a depth of 45 feet of seawater (fsw) (modified U.S. Navy Treatment Table 9). The chamber was compressed over a 10-minute time interval representing a 4.5 fsw/minute uniform rate of compression. This 4.5-fsw/minute linear rate (slope) of compression rate was maintained throughout the total 10-minute time interval of treatment and will be used as a baseline compression rate to compare all other compression schedules [total compression time interval/compression rates (slopes)]. The investigators will prospectively collect data on patient-treatment group exposures after formalizing four different compression schedules each including a unique combination of compression rate (slope) and time intervals of compression. This was similar to the Phase I study.

Data will be collected prospectively on all patients recruited and receiving treatment from February 11, 2019, and February 10, 2020, and combined with the data obtained in our Phase I trial collected from September 8, 2014 to September 8, 2016. This Phase II study defines the unit of observations as a multiplace patient-treatment group exposure rather than individual patient treatment exposures. This approach was considered appropriate as a treatment stop or hold in a multiplace chamber affects all other patient occupants in the same treatment group exposure.

To mitigate the risk of confounding, only the first stop will be used as the stop or hold indicator for that particular patient-treatment group exposure. Data will be collected on the patient(s) experiencing the stop or hold. All patients will undergo pre-treatment video otoscopy with baseline tympanic membrane (TM) photos and video of TM motion documenting the patients ability to equalize. This is used to assess potential Eustachian tube patency and proper equalization performance to help exclude individual patient technique as a confounding variable. Photos will be repeated at the end of treatment on any patient(s) complaining of symptoms referable to ETD/MEB that require a stop during compression.

Multiple stops for the same patient on the same treatment will not be considered. Only the first compression stop or hold during each treatment exposure will be recorded or assigned as a patient-treatment stop representing that particular patient-treatment group exposure. Compression stops will be made when any patient experiences difficulty equalizing (requests a stop or complains of ear discomfort of any type).

Repeat video otoscopy will be conducted on all patients complaining of symptoms referable to ETD or MEB to objectively document the grade of barotrauma at the end of the treatment. The OGS system will be used to record the severity of the ETD or MEB. The depth of the stop, the treatment number for that particular patient, and the actions taken to alleviate the symptoms during equalization will be recorded.

The depth of the compression stop will be recorded in feet of seawater (fsw) as will be the ascent (fsw) required for the patient to clear the middle ear pressure and relieve the symptoms. The patients symptoms must be resolved, rendering the patient asymptomatic and able to continue the treatment compression profile. All team members (physicians, nurses, and technicians) present and working on the day of the exposure, are responsible for viewing the patients pre and post tympanic membrane photos and determining the grade of barotrauma using the OGS criteria.

All stops were categorized under the respective compression protocol used for that particular patient-treatment group exposure. Data will then compared using both descriptive and inferential statistical analysis including the risk difference, odds ratio (OR), two-tailed Chi Square analysis using α=0.05, and outcomes will be studied separately in a logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria: Any patient meeting the indications for hyperbaric oxygen treatment.

-

Exclusion Criteria: Any patient with absolute contraindications to hyperbaric oxygen treatment, chronic bilateral perforation of the tympanic membrane or prior bilateral myringotomy tube placement.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Compression stops or holds during the compression phase of hyperbaric oxygen treatments | Patients are assessed during each hyperbaric chamber compression until reaching treatment pressure/depth daily throughout the entire treatment course that varies based on diagnosis over 4-12 weeks
  Hyperbaric oxygen treatment (HBOT) protocols include a compression phase. Pressure is increased until final treatment pressure is achieved. Pressure changes vary between 14.7 psi to 35 psi. Patients experience symptoms of pain or pressure in the middle ear space because they cannot clear middle ear pressure. Pressure symptoms may be time and/or slope related. Using varying rates of pressure may decrease discomfort related to clearing middle ear pressure; Eustachian tube dysfunction (ETD) and middle ear barotrauma (MEB), the most common adverse effects of HBOT. The authors believe a slower rate or slope of compression may decrease the occurrence of stops and decrease the incidence of ETD and MEB during HBOT. Decreasing rate of compression may further mitigate risk and decrease the incidence of symptomatic ETD and MEB.
Assessing the severity of Eustachian tube dysfunction and middle ear barotrauma after using various compression rates and slopes of compression during hyperbaric oxygen treatment via direct video otoscopy | Patients are assessed during each hyperbaric chamber compression until reaching treatment pressure/depth daily throughout the entire treatment course that varies based on diagnosis over 4-12 weeks
  Photo otoscopy and the severity of eustachian tub dysfunction and/or middle ear barotrauma will be defined using the O'Neill Grading System when a patient experiences a stop or hold during the compression phase of hyperbaric oxygen treatment.
  O'Neill Grading System:
  0 = Symptoms of Eustachian tube dysfunction with no objective signs of barotrauma on otoscopy
  1. = Objective evidence of increased erythema, air trapping or serous/serosanguinous effusion
  2. = Any frank bleeding in the middle ear space, tympanic membrane or external ear canal or perforation

CONTACTS AND LOCATIONS:
Overall Officials: Owen J O'Neill, MD, MPH, Principal Investigator — Phelps Hospital Northwell Health
Locations (1):
- Phelps Hospital Northwell Health, Sleepy Hollow, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Would consider if other researchers are studying similar research question and interested in collaboration.
Supporting Information: Study Protocol, CSR
Time Frame: Post publication
Access Criteria: Contact Primary Investgators by Email

REFERENCES:
- [Background] 1. Beuerlein M, Nelson RN, DB W. Inner and middle ear hyperbaric oxygen induced barotrauma. The Laryngoscope. 1997;107(10):1350-6. 2. EM C. Side effects of hyperbaric oxygen therapy. Undersea & Hyperbaric Medicine : Journal of the Undersea and Hyperbaric Medical Society, Inc. 2014;41(3):253-7. 3. Heyboer M, Wojcik SM, Grant WD, Chambers P, Jennings S, P A. Middle ear barotrauma in hyperbaric oxygen therapy. Undersea & Hyperbaric Medicine Journal of the Undersea and Hyperbaric Medical Society, Inc, . 2014;41(5):393-7. 4. Lima MA, Farage L, Cury MC, FJ B. Update on middle ear barotrauma after hyperbaric oxygen therapy-insights on pathophysiology. International Archives of Otorhinolaryngology. 2014;18(2):204-9. 5. Ng AWA, Muller R, J O. Incidence of middle ear barotrauma in staged versus linear chamber compression during hyperbaric oxygen therapy: a double blinded, randomized controlled trial. Undersea Hyperb Med: Journal of the Undersea and Hyperbaric Medical Society, Inc. 2017;44(2):101-7. 6. Plafki C, Peters P, Almeling M, Welslau W, R B. Complications and side effects of hyperbaric oxygen therapy. Aviation, Space, and Environmental Medicine. 2000;71(2):119-24. 7. Toklu AS, Shupak A, Yildiz S, Aktas S, Ertracht O, Ay H, et al. Aural barotrauma in submarine escape: is mastoid pneumatization of significance? The Laryngoscope. 2005; 115(7):1305-9. 8. Vahidova D, Sen P, Papesch M, Zein-Sanchez MP, PH M. Does the slow compression technique of hyperbaric oxygen therapy decrease the incidence of middle ear barotrauma? J Laryngol Otol. 2006;120(6):446-9. 9. Varughese L, O'Neill OJ, Marker J, Smykowski E, Dayya D. The Effect of Compression Rate and Slope on the Incidence of Symptomatic Eustachian Tube Dysfunction Leading to Middle Ear Barotrauma: A Phase 1 Prospective Study. Undersea & Hyperbaric Med: Journal of the Undersea and Hyperbaric Medical Society, Inc. 2019;46(2):95-100. 10. AA B. Diving medicine. American Journal of Respiratory and Critical Care Medicine. 2014;189(12):1479-86. 11. Fitzpatrick DT, Franck BA, Mason KT, SG S. Risk factors for symptomatic otic and sinus barotrauma in a multiplace hyperbaric chamber. Undersea & Hyperbaric Medicine : Journal of the Undersea and Hyperbaric Medical Society, Inc. 1999;26(4):243-7. 12. Goplen FK, Gronning M, Aasen T, SHG N. Vestibular effects of diving -- a 6-year prospective study. . Occup Med 2010;60(1):43-8. 13. Hadanny A., Meir O, Bechor Y., Fishlev G, Bergan J, S E. The safety of hyperbaric oxygen treatment--retrospective analysis in 2,334 patients. Undersea & Hyperbaric Medicine: Journal of the Undersea and Hyperbaric Medical Society, Inc. 2016;43(2):113-22. 14. Mozdzanowski C, GA P. Peripheral neuropathy may increase the risk for asymptomatic otic barotrauma during hyperbaric oxygen therapy: Research report. Undersea & Hyperbaric Medicine: Journal of the Undersea and Hyperbaric Medical Society, Inc. 2014;41(4):267-72. 15. RW S. Controlling the rate of middle ear barotrauma: An editorial perspective. Undersea & Hyperbaric Medicine : Journal of the Undersea and Hyperbaric Medical Society, Inc. 2014;41(5):355-6. 16. O'Neill OJ, ED W. The O'Neill grading system for evaluation of the tympanic membrane: A practical approach for clinical hyperbaric patients. Undersea & Hyperbaric Medicine : Journal of the Undersea and Hyperbaric Medical Society, Inc. 2015;42(3):265-71. 17. Mozdzanowski C, GA P. Peripheral Neuropathy May Increase the Risk for Asymptomatic Otic Barotrauma During Hyperbaric Oxygen Therapy: Research Report. Undersea and Hyperbaric Medicine Journal of Undersea and Hyperbaric Medical Society. 2014;41(4):267-72. 18. Nasole E, Zanon V, Marcolin P, G B. Middle Ear Barotrauma During Hyperbaric Oxyeg Therapy; A Review of Occurrences in 5962 Patients. Undersea & Hyperbaric Med: Journal of the Undersea and Hyperbaric Medical Society. 2019;46(2):101-6.
- [Derived] O'Neill OJ, Dayya D, Varughese L, Marker JA, Perez L, Dayya M. The effect of total compression time and rate (slope) of compression on the incidence of symptomatic Eustachian tube dysfunction and middle ear barotrauma: a Phase II prospective study. Undersea Hyperb Med. 2021 Third Quarter;48(3):209-219. PMID 34390625